CLINICAL TRIAL: NCT06872463
Title: Brain Immunoactivation in Drug-Naive Patients with First Episode Schizophrenia
Brief Title: Karolinska Schizophrenia Project
Acronym: KaSP
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Centre for Psychiatry Research, Region Stockholm, Sweden (Unknown)
Responsible Party: Principal Investigator, Carl Sellgren, Associate Professor Carl Sellgren Majkowitz, Karolinska Institutet
Other Study IDs: 2010/879-31/1
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia and Disorders with Psychotic Features
Keywords: Psychosis; Psychotic disorders; Schizophrenia
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid (CSF), whole blood, fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- First Episode Psychosis (FEP): Diagnosis of psychotic disorder according to the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV), where anti-psychotic medication was initiated less than four weeks prior to inclusion.
- Healthy Control (HC): Age and sex matched individuals

SUMMARY:
KaSP is a multimodal observational study with the goal of clarifying underlying mechanisms that cause psychotic disorders, such as schizophrenia. Participants with psychotic symptoms are recruited early after first contact with health care, within 4 weeks of starting anti-psychotic medication, and are compared to controls without psychiatric diagnoses on several measures.

DETAILED DESCRIPTION:
KaSP aims to recruit 120 patients sparsely medicated or drug-naive first episode psychosis (FEP) individuals, along with 80 healthy controls.

Participants undergo the following assessments and measurements:

* Clinical assessment
* Cognitive testing
* Lab results from cerebrospinal fluid, blood, urine, saliva and skin biopsy
* Brain imaging using Magnetic Resonance Imaging (MRI) and Positron Emission Tomography (PET)
* Pre-Pulse Inhibition (PPI) (a test to evaluate the startle response)
* Measures of arterial stiffness and amount of vascular narrowing

Participants with psychosis are invited back for repeat measurements at 1,5 and 5 years after study enrollment. Controls may be invited back at 1,5 years for repeat of some of the assessments.

ELIGIBILITY:
Inclusion Criteria:

For FEP:

* Diagnosis as assessed using DSM-IV of one of the following: schizophrenia, schizophreniform psychosis, psychosis not otherwise specified (NOS), brief psychosis, schizoaffective syndrome, delusional disorder
* First exposure to anti-psychotic medication less than 4 weeks prior to inclusion

Exclusion Criteria:

For FEP:

- Other dominant psychiatric illness deemed to be related to current psychotic symptoms

For HC:

* A history of diagnosis of a major psychiatric disorder, including substance use disorders.
* Family history of psychotic disorders in first degree relatives.

For all:

* Evidence based on medical history, clinical signs, MRI or laboratory tests of clinically significant somatic disorder, or previous disorder with brain engagement (e.g. tumour, neuroinflammatory disease, epilepsy) or significant brain trauma.
* Exposure to an effective radiation dose of 25 mSv during the past year.
* Pregnancy, lactating or breastfeeding (women).
* Meets diagnostic criteria of substance use disorder (excluding nicotine dependence) as assessed using DSM-IV or as determined using repeated positive urine screens during the course of the study.
* Metallic object in the eye, or ferro/electromagnetic implants. History of claustrophobic anxiety during MRI.
* Symptoms of severe bacterial, fungal, or viral infection (including upper respiratory tract infection), with systemic effects as detected by e.g. fever, within 7 days prior to inclusion.
* Treatment with any antihemostatic medication within 2 weeks of lumbar puncture and arterial line placement of either the baseline or 1 year follow-up.
* Blood donation (1 unit or more) within 90 days prior to Screening, plasma donation from 1 week prior to Screening, and platelet donation from 6 weeks prior to inclusion.
* Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the participant unsuitable for enrollment. This may include very high symptom severity or signs of aggressiveness and hostility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: FEP are recruited from psychiatry clinics in the greater Stockholm area. HC are recruited by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Kynurenic acid (KYNA) in FEP compared to HC | Baseline measure
  KYNA are measured in CSF and blood samples
Cytokines in FEP compared to HC | Baseline measure
  Cytokines are measured in CSF and blood samples
Microglial activation in FEP compared to HC | Baseline measure
  Group comparison of binding of the PET ligand [11C]PBR-28
Dopamine receptors in FEP compared to HC | Baseline measure
  Group comparison of binding of the PET-ligand [11C]FLB457
Infectious risk factors in FEP and subsequent relation to clinical outcome | Registry data in childhood, measurement at baseline, registry data through study completion (with an expected average of 7 years of follow up)
  Registry data on previous infections, along with infectious agents measured in CSF and blood. Long term clinical outcome is measured through registry data, by drug-dispensation as well as in-and outpatient care for both somatic and psychiatric disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- SLSO Psykiatri Stockholm in collaboration w Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://ki.se/en/research/research-areas-centres-and-networks/research-groups/applied-developmental-neurobiology-carl-sellgren-research-group#tab-the-karolinska-schizophrenia-project-kasp-